CLINICAL TRIAL: NCT01272297
Title: The Effect of Low Intensity Shock Wave Therapy in Severe ED Patients Not Responding to Oral Medication
Brief Title: The Effect of Low Intensity Shock Wave Therapy for ED in PDE5i Non Responders
Acronym: LI-ESWT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Medispec (Industry)
Responsible Party: Principal Investigator, i_gruenwald, MD, Rambam Health Care Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: shock wave III
Record Dates: First submitted 2010-12-14; First posted 2011-01-07 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Erectile Dysfunction
Keywords: LI-ESWT; Erectile Dysfunction; Non PDE5 inhibitor responders; Shock wave
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LI-ESWT (Experimental): Low intensity shock wave treatment- 12 sessions
  Interventions: Device: LI-ESWT

INTERVENTIONS:
Device: LI-ESWT — Low intensity shock wave treatment - 12 sessions
  Other Names: Omnispec model ED1000

SUMMARY:
Low Intensity Shock Wave Therapy (LI-ESWT) was shown to have a beneficial effect on ED patients responding to PDE5i's. This study aimed to determine the capability of swt to convert PDE5 inhibitor non responders to sexually functioning males under PDE5i therapy.

DETAILED DESCRIPTION:
We included severe ED patients (60% diabetic, 85% with cardiovascular disease) that failed to respond to PDE5i therapy, who scored 0-2 on the rigidity scale (RS) during PDE5i therapy.Treatment included 2 sessions/week for 3 weeks, repeated after a 3-week no-treatment interval. At each session LI-ESWT was applied on the penile shaft and crus for 3 minutes in 5 different penile anatomical sites (intensity of 0.09 mj/mm2, 300 shocks/site). One-month after end of treatment the same baseline assessment was repeated. An active PDE5i medication regime was then provided and final erectile function was reassessed. Main endpoints for success were changes in RS and in the International Index of Erectile Function (IIEF-ED) Domain score. We found that LI-ESWT can effectively treat severe ED patients who failed PDE5i therapy. This study further emphasises the physiological effect that LI-ESWT can have on the erectile mechanism.

ELIGIBILITY:
Inclusion Criteria:

* ED of more than 6 months
* Rigidity score ≤ 2 during PDE5i therapy
* Stable heterosexual relationship for more than 3 months
* Patients need to know and to agree that the study protocol does not allow any PDE5I therapy till week 13 .

Exclusion Criteria:

* Prior surgery or radiotherapy in pelvic region
* Any unstable, psychiatric, spinal cord injury and penile anatomical abnormalities
* Clinically significant chronic hematological disease
* Anti-androgens, oral or injectable androgens
* Cardiovascular conditions that prevent sexual activity

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
IIEF-ED Domain score | 17 weeks after first visit
  Change of 5 points and above in IIEF-ED Domain score

SECONDARY OUTCOMES:
rigidity scale | 17 weeks from visit 1
  a change to 3 or 4 points in the rigidty scale

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Vardi, Prof, Principal Investigator — Rambam Health Care Campus; Ilan Gruenwald, MD, Study Director — Rambam Health Care Campus; Boaz Appel, MD, Study Director — Rambam Health Care Campus; Ezra Gerber, RN, Study Director — Rambam Health Care Campus; Yaron Ofer, MD, Study Director — Rambam Health Care Campus; Omar Massarwa, RN, Study Director — Rambam Health Care Campus